CLINICAL TRIAL: NCT02558010
Title: Perioperative Methadone Use to Decrease Opioid Requirement in Pediatric Spinal Fusion Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Keri Hainsworth, Associate Professor, Medical College of Wisconsin
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CHW-Methadone-001
Record Dates: First submitted 2015-02-13; First posted 2015-09-23 (Estimated); Results first posted 2023-04-27 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Scoliosis; Pain
Keywords: Methadone; Gabapentin; Postoperative Pain; Posterior Spinal Fusion; Pediatric
MeSH Terms: conditions — Scoliosis; Pain; Pain, Postoperative | interventions — Methadone; Saline Solution; Fluoridation; Morphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Methadone Group (Experimental): Patients will receive a total of 0.2mg/kg IV methadone intraoperative (0.1mg / kg preincision and 0.1mg/kg prior to emergence) with a maximum dosing of 20 mg.
  Interventions: Drug: Methadone; Drug: Morphine
- Control Group (Active Comparator): Patient will receive normal saline placebo initially, then morphine prior to emergence.
  Interventions: Other: Normal Saline; Drug: Morphine

INTERVENTIONS:
Drug: Methadone — Perioperative IV methadone to be given
  Other Names: generic methadone
  Arms: Methadone Group
Other: Normal Saline — control arm
  Other Names: salt water
  Arms: Control Group
Drug: Morphine — Both groups will receive morphine via Patient-Controlled Analgesia (PCA) pump.
  Other Names: Duramorph

SUMMARY:
Acute pain management following major surgical procedures in pediatric patients continues to be a challenge, especially after extensive posterior spine fusions.

Spine surgery is particularly traumatic, initiating pain in both peripheral and central pathways. While the standard management of post-surgical pain involves a multimodal approach, opioids provide the predominant benefit. However, opioid use is associated with many adverse effects, including nausea, constipation, and pruritus. Perioperative methadone may decrease total opioid consumption and adverse effects as well as improve satisfaction with pain management after scoliosis repair.

DETAILED DESCRIPTION:
This study is a double blind comparison, evaluating the benefits of intraoperative methadone in extensive posterior spine fusion surgery for idiopathic scoliosis. Methadone 0.2 mg/kg will be given to the treatment group. Postoperative evaluation for narcotic use, pain control, and adverse effects will be compared to a standard treatment approach used at Children's Hospital of Wisconsin.

ELIGIBILITY:
Inclusion Criteria:

* Age 10-18 years
* Idiopathic scoliosis
* Fusion levels planned for 10 or greater
* English speaking
* American Society of Anesthesiology (ASA) class 1 - 3

Exclusion Criteria:

* Current narcotic use / History of substance use disorder
* Morphine, hydromorphone or methadone allergies
* Pregnancy
* Seizure disorders
* Bleeding disorders
* Neuromuscular scoliosis
* History of renal or hepatic disease
* Long QT syndrome
* Obstructive sleep apnea
* Body mass index > 40
* Inability to tolerate standard analgesic medications (gabapentin, ketorolac, acetaminophen)
* Non-English speaking

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 58 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2023-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Weisman, MD, Study Chair — Children's Hospital and Health System Foundation, Wisconsin; Roger A Fons, MD, Principal Investigator — Children's Hospital and Health System Foundation, Wisconsin
Locations (1):
- Children's Wisconsin, Milwaukee, Wisconsin, United States

REFERENCES:
- [Background] Berde CB, Beyer JE, Bournaki MC, Levin CR, Sethna NF. Comparison of morphine and methadone for prevention of postoperative pain in 3- to 7-year-old children. J Pediatr. 1991 Jul;119(1 Pt 1):136-41. doi: 10.1016/s0022-3476(05)81054-6. PMID 2066846
- [Background] Gottschalk A, Durieux ME, Nemergut EC. Intraoperative methadone improves postoperative pain control in patients undergoing complex spine surgery. Anesth Analg. 2011 Jan;112(1):218-23. doi: 10.1213/ANE.0b013e3181d8a095. Epub 2010 Apr 24. PMID 20418538
- [Background] Rusy LM, Hainsworth KR, Nelson TJ, Czarnecki ML, Tassone JC, Thometz JG, Lyon RM, Berens RJ, Weisman SJ. Gabapentin use in pediatric spinal fusion patients: a randomized, double-blind, controlled trial. Anesth Analg. 2010 May 1;110(5):1393-8. doi: 10.1213/ANE.0b013e3181d41dc2. PMID 20418301
- [Background] Sharma A, Tallchief D, Blood J, Kim T, London A, Kharasch ED. Perioperative pharmacokinetics of methadone in adolescents. Anesthesiology. 2011 Dec;115(6):1153-61. doi: 10.1097/ALN.0b013e318238fec5. PMID 22037641

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Methadone Group | Control Group
Started | 30 | 28
Completed | 25 | 22
Not Completed | 5 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Methadone Group | Control Group | Total
Number analyzed (Participants) | 25 | 22 | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.0 (1.8) | 14.6 (2.3) | 14.81 (2.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 17 | 38
  Male | 4 | 5 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 24 | 20 | 44
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 2 | 6
  White | 20 | 18 | 38
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 25 | 22 | 47

OUTCOME MEASURES:

1. Primary Outcome: Post-operative Opioid Consumption (mg/kg)
Description: Total amount of opioids consumed during the first 72 hours after surgery.
Time Frame: 72 hours
Population: All participants allocated to study groups, and received the intervention.
Measure: Median (Inter-Quartile Range); unit: mg/kg
Arm/Group | Methadone Group | Control Group
Number analyzed (Participants) | 25 | 22
mg/kg | 0.267 [0.119 to 0.451] | 0.340 [0.168 to 0.607]
Statistical Analysis 1: Comparison: Methadone Group vs Control Group; Test type: Superiority; p < 0.05, Mixed Models Analysis — The p-value was calculated, and does not indicate the threshold for statistical significance

ADVERSE EVENTS:
Time Frame: Three post-operative days.
Description: Data represent the number of patients treated for each side effect, collapsed across post-operative days.
Arm/Group | Methadone Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/22
Other Adverse Events (participants affected / at risk) | 1/25 | 0/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Methadone Group (N=25) | Control Group (N=22)
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-12): https://cdn.clinicaltrials.gov/large-docs/10/NCT02558010/Prot_SAP_001.pdf